CLINICAL TRIAL: NCT03654911
Title: Sustainable Method for Alzheimer's Prediction in Mild Cognitive Impairment: EEG Connectivity and Graph Theory Combined With ApoE Testing.
Brief Title: Sustainable Method for Alzheimer's Prediction
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Paolo Maria Rossini, Full Professor, Catholic University of the Sacred Heart
Other Study IDs: ROSSINI_MSD_ID1764
Record Dates: First submitted 2018-07-10; First posted 2018-08-31 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease; Amnestic-Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease | interventions — Electroencephalography; Apolipoproteins E

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aMCI subjects: EEG recording, ApoE testing
  Interventions: Diagnostic Test: EEG; Genetic: ApoE

INTERVENTIONS:
Diagnostic Test: EEG — EEG
Genetic: ApoE — ApoE

SUMMARY:
This is an observational study with the aim of validating, in a consistent population sample, with appropriate follow-up, whether EEG connectivity analysis combined with the neuropsychological evaluation and ApoE genotype testing in aMCI could be of help in early identification of converted aMCI as a first-line screening method in order to intercept early those subjects with a high risk for rapid progression to AD.

DETAILED DESCRIPTION:
Primary aim of the present project is to investigate the dynamic connectivity among brain centers by using a mathematical (Small World) approach to the analysis of EEG-related neural networks. The aim is to provide reliable discrimination of amnesic-Mild Cognitive Impairment (a MCI) subjects who, on individual basis, will rapidly convert to Alzheimer Disease (AD) after a relatively brief follow-up. Moreover, keeping in mind that the epsilon-4 allele of the ApoE gene is a genetically determined risk factor for pathogenesis of late-onset AD, a secondary endpoint is introduced to investigate whether the EEG connectivity markers together with a genetically determined risk of dementia as represented by ApoE testing can reach higher sensitivity/specificity for early discrimination of MCI converting to AD

ELIGIBILITY:
Exclusion criteria for AD will be:

* frontotemporal dementia;
* behavioural variant of frontotemporal dementia;
* vascular dementia;
* extra-pyramidal syndromes;
* reversible dementias (including pseudodementia of depression);
* Lewy body dementia.

The exclusion criteria for aMCI will be:

* mild AD, as diagnosed by standard protocols including National Institute on Aging-Alzheimer's Association workgroups (McKhann et al. 2011);
* evidence (including magnetic resonance imaging -MRI procedures) of concomitant dementia such as frontotemporal, vascular and reversible dementias (including pseudo-depressive dementia), marked fluctuations in cognitive performance compatible with Lewy body dementia and/or features of mixed dementias;
* evidence of concomitant extrapyramidal symptoms;
* clinical and indirect evidence of depression as revealed by the Geriatric Depression Scale GDS (Yesavage et al. 1982); scores lower than 14 (no depression);
* other psychiatric diseases, epilepsy, drug addiction, alcohol dependence, use of neuro/psychoactive drugs including acetylcholinesterase inhibitors;
* current or previous uncontrolled or complicated systemic diseases (including diabetes mellitus) or traumatic brain injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants 150 aMCI will be recruited (including 90 already available EEG and clinical data recordings) in order to obtain two homogeneous sub-groups according to the clinical follow-up, classifying them as converted to AD or stable aMCI after a 12 to 24 months period from the time of baseline EEG recording.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Biomarkers: EEG | 2 years
  EEG recording will be performed at rest, with closed eyes from routine electrode scalp positions according to the International 10-20 system. Functional connectivity analysis will be performed using eLORETA evaluating intracortical Lagged Linear Coherence. Weighted and undirected networks will be built from the above measure. Small World parameter is a dimentionless number that will be assessed as Biomarker of brain connectivity networks, since it measures the balance between local connectedness and the global integration of a network, representing brain network organization. Small world index will be computed in the seven EEG frequency bands delta (2-4 Hz), theta (4-8 Hz), alpha 1 (8-10.5 Hz), alpha 2 (10.5-13 Hz), beta 1 (13-20 Hz), beta 2 (20-30 Hz) and gamma (30-45 Hz) (Vecchio et al., 2018 doi: 10.1002/ana.25289)
Biomarker: ApoE4 | 2 years
  It will be evaluated the allele of the Apo-E gene as biomarker for the pathogenesis of late-onset and sporadic AD. The Apo-E test provides a dimentionless value represented by the type of the allele (ε2, ε3,ε4).

SECONDARY OUTCOMES:
Biomarker: Accuracy of digital classifier | 2 years
  Secondary endpoint will be to investigate whether EEG connectivity markers (small world ) along with genetically determined risk-indicators for dementia, as represented by Apo-E testing can reach a greater sensitivity, specificity and accuracy for a digital classifier (i.e. an algorithm that solve the problem of identifying to which of a set of categories a new observation belongs) able to predict the MCI conversion to AD. The accuracy value is dimentionless number represented by a percentual value and it is the biomarker for the ability of the classifier for the early identification of AD (Vecchio F. et al., 2018 doi: 10.1002/ana.25289)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico A.Gemelli IRCCS, Università Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vecchio F, Miraglia F, Iberite F, Lacidogna G, Guglielmi V, Marra C, Pasqualetti P, Tiziano FD, Rossini PM. Sustainable method for Alzheimer dementia prediction in mild cognitive impairment: Electroencephalographic connectivity and graph theory combined with apolipoprotein E. Ann Neurol. 2018 Aug;84(2):302-314. doi: 10.1002/ana.25289. Epub 2018 Aug 25. PMID 30014515